CLINICAL TRIAL: NCT01745068
Title: Partnership for Applied Research in Fracture Prevention Programs for the Elderly
Acronym: OPTI-FRAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ministere de la Sante et des Services Sociaux (Other); Merck Sharp & Dohme LLC (Industry); Novartis (Industry); Amgen (Industry); CSSS-IUGS Estrie (Unknown)
Responsible Party: Principal Investigator, Isabelle Gaboury, Assistant professor, Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIHR grant # 267395
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Osteoporosis With Current Fragility Fracture
Keywords: fragility fracture; osteoporosis; fall prevention; integrated program; interorganizational collaboration; Canada; controlled clinical trial; evaluation
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention)
- Integrated program (Experimental): Participants will be involved in an integrated interorganisational fragility fracture prevention program, which combines both post-fracture management as well as fall prevention strategies. The intervention will last up to 18 months.
  Interventions: Other: Integrated program

INTERVENTIONS:
Other: Integrated program — Each participant's primary care physician will receive written information containing a presumed osteoporosis diagnosis, investigations to be performed, correct interpretation of any bone densitometry results in the context of a fragility fracture, and treatment options. The study coordinator will be responsible for orienting the participant to an appropriate local fall prevention program.
  Arms: Integrated program

SUMMARY:
During their lifetime, approximately 50% of Canadian women and 30% of Canadian men will experience at least one fracture due to bone fragility (FF). Evidence is growing regarding prevention programs' effectiveness to prevent falls, but prevention of fractures through fall prevention programs has enjoyed limited success. Falls prevention programs and post-fracture screening programs leading to pharmacological treatment are very different strategies, with a shared ultimate goal. Coordination between those who repair fractures and those who manage the patient to prevent the next fracture is critical. The overarching aim of this proposal is to generate evidence-based knowledge about the effectiveness and cost-effectiveness of an integrated FF prevention program, as well as a portrait of the barriers and facilitating factors for such programs. More specifically, the objectives are: 1) to combine existing fall prevention and post-fracture management programs in the province of Quebec into integrated FF prevention programs; 2) to compare the performance of these integrated programs to control sites, using a pragmatic study design; 3) to identify barriers as well as factors that improve effectiveness across different implementation milieu; and 4) to develop and engage in active knowledge transfer activities in Quebec regions where integrated FF prevention programs are neither adequately nor successfully implemented. Drawing upon the literature on integrated healthcare, fall and fracture prevention, we hypothesize that an integrated FF program can reduce the risk of a subsequent fracture by at least 30% in the population of interest. The proposed team is poised to develop new interdisciplinary collaborations among healthcare practitioners and decision makers involved in the prevention of FFs. The program is built upon existing healthcare and structures and programs and in turn, will truly measure the effectiveness of an integrated FF prevention program. The results will ultimately lead to improvements in the existing knowledge base, address policy-relevant and health systems problems, and assist in the design and implementation of FFs prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age and over
* must have a primary care physician
* must be able to follow simple instructions
* must have sustained a fragility fracture within three months of the recruitment date.

Exclusion Criteria:

* severe kidney insufficiency (grade 4 or 5)
* advanced stage of cancer
* fracture to sites not commonly associated with osteoporosis such as toe, finger, hand, foot, ankle, patella, head, and cervical spine.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2013-01; Primary Completion 2016-11 (Actual); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of secondary fragility fracture | 18 months post recruitment

SECONDARY OUTCOMES:
Initiation of osteoporosis treatment by the primary care physician | At 6, 12, 18, and 60 months post recruitment
  Osteoporosis treatment includes bisphosphonates or other effective osteoporosis drugs.
Compliance with osteoporosis treatment. | At 6, 12, 18, and 60 months post recruitment
  The data collected from the participant will be validated with the participant's pharmacist through the medication possession ratio. The medication possession ratio is measured from the first to the last prescription, with the denominator being the duration from index to the exhaustion of the last prescription and the numerator being the days supplied over that period from first to last prescription and the numerator being the total number of days in the interval.
Time to first fall event | Within the first 18 months post recruitment
Incidence of secondary fragility fractures. | At 24, 36, 48 and 60 months post recruitment
Number of clinically significant fall events. | At 18, 24, 36, 48 and 60 months post recruitment
Fall-related hospitalizations | At 18, 24, 36, 48 and 60 months post recruitment
  Fall-related hospitalizations will be recorded in the participant diary and at each telephone follow-up, and validated with the participant's hospital records.
Fragility fracture-related death | At 18, 24, 36, 48 and 60 months post recruitment
  Fragility fracture-related death will be confirmed from a provincial administrative database (Regie de l'assurance maladie du Quebec - RAMQ).
Participants' quality of life | At 18, 24, 36, 48 and 60 months post recruitment
  Euro-QOL
Practice of physical activities | At 6, 12, 18, 24, 36, 48 and 60 months post recruitment
  CHAMPS
Fragility fracture-related costs | At 18 and 60 months post recruitment
  Medical costs from the participant's hospital record include: medical assessment, prescription and non-prescription drugs; and resource use related to the management of the fragility fracture and/or long-term complications, including hospitalization. As well, lost days of work, annual income (if the participant is in the labour force), travel to the hospital and/or rehabilitation facilities, parking, and out-of-pocket expenses for drugs and rehabilitation devices (e.g. splint) will be compiled. Protocol-driven costs will be excluded, with the exception of the costs related to the participants' fall prevention program.
Admission to a long-term care facility | At 18, 24, 36, 48 and 60 months post recruitment
Participants' perceptions of care integration | At 12 months post intervention
  All participants' perceptions of care integration will be captured 12 months after the beginning of the intervention period, or following an early withdrawal from the study.
Intervention participant's satisfaction with the fragility fracture prevention program | At 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Gaboury, PhD, Principal Investigator — Université de Sherbrooke; Hélène Corriveau, PhD pht, Principal Investigator — Université de Sherbrooke
Locations (10):
- Canada (10):
  - Centre hospitalier Hôtel-Dieu d'Amos, Amos, Quebec
  - CSSS du Roché Percé (Centre hospitalier de Chandler), Chandler, Quebec
  - Hôpital de Hull, Gatineau, Quebec
  - Hôpital Charles Lemoyne, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Hôpital Jean-Talon, Montreal, Quebec
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre hospitalier régional de Lanaudière, Saint-Charles-Borromée, Quebec
  - CSSS de St-Jérôme (Hôpital régional de St-Jérôme), Saint-Jérôme, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Gaboury I, Corriveau H, Boire G, Cabana F, Beaulieu MC, Dagenais P, Gosselin S, Bogoch E, Rochette M, Filiatrault J, Laforest S, Jean S, Fansi A, Theriault D, Burnand B. Partnership for fragility bone fracture care provision and prevention program (P4Bones): study protocol for a secondary fracture prevention pragmatic controlled trial. Implement Sci. 2013 Jan 24;8:10. doi: 10.1186/1748-5908-8-10. PMID 23343392